CLINICAL TRIAL: NCT07122791
Title: Investigation of the Effects of Tele-rehabilitation-based Motor Imagery Training on Kyphotic Angle, Pain, Depression, and Quality of Life in Individuals With Posture Disorders.
Brief Title: Investigation of the Effectiveness of Tele-rehabilitation Based Motor Imagery Training in Individuals With Posture Disorders.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Emrah Zirek, Assistant Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BingolUni
Record Dates: First submitted 2024-10-02; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2023-10

CONDITIONS: Posture; Kyphosis; Muscle Cramps; Thoracic Vertebrae
Keywords: Telerehabilitation; Manipulation, Orthopedic; Posture
MeSH Terms: conditions — Kyphosis; Muscle Cramp

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Home Exercise Program Group (Experimental): Home exercise program that includes strengthening and stretching
  Interventions: Other: Home Exercise Group
- Group 2: Home Exercise Program + Motor Imagery Training (Experimental): Motor imagery training, in addition to the home exercise program, was applied twice a week for 6 weeks via tele-rehabilitation under the supervision of a physiotherapist.
  Interventions: Other: Home Exercise Group

INTERVENTIONS:
Other: Home Exercise Group — In addition to the exercise program, Group 2 will receive motor imagery training. This will be carried out using the telerehabilitation method, under the supervision of a physiotherapist, and will be delivered twice a week for six weeks. A text containing posture exercises will be prepared by the physiotherapist for motor imagery training. The motor imagery text will be updated as the home exercise program is completed. The content of the motor imagery program will consist of 5 minutes of relaxation and 15 minutes of imagery training. Relaxation training will include relaxation and breathing exercises. After relaxation training, the patient will be asked to stand up with his eyes closed in a safe environment where he feels comfortable, and then a text containing posture exercises prepared by the physiotherapist for motor imagery will be read. The patient will be asked to perform the exercise by imagining it in his mind without moving his body.

SUMMARY:
Objective: Kyphosis is one of the most common postural problems. It is defined as a thoracic curvature that exceeds normal limits. The Cobb angle, also known as the kyphosis index, can be used to determine the degree of this curvature. Motor imagery (MI) is defined as visualising movement in the mind without actually moving. Studies have shown that similar brain regions are activated during motor imagery and actual movement.

regions are activated during motor imagery and actual movement. Most of the information about motor imagery training has been obtained from studies of stroke patients, and the physical effects of motor imagery training have been examined in these studies.

However, there has been no study in which motor imagery, which is mostly performed by neurological stroke groups or athletes, is used for treatment of postural disorders. In this context, this study aims to examine the effect of tele-rehabilitation-based motor imagery training on kyphotic angle, pain, depression and quality of life in individuals with posture disorders.

Materials and methods: Young adults with postural kyphosis who are studying at Istanbul University-Cerrahpaşa Faculty of Health Sciences will be included in the randomised controlled, double-blind, prospective study.

of Health Sciences and who volunteered to participate in the study, will be included in the randomised controlled, double-blind, prospective study.

Participants will be randomly divided into two groups: an exercise group (Group 1) and an exercise + motor imagery group (Group 2).

The presence of kyphosis in participants will be evaluated by measuring the Flexruler kyphosis index and wall-occiput distance.

Posture will be evaluated using the New York Posture Analysis and pain using a visual pain scale. Depression will be assessed using the Beck Depression Scale.

assessment will be evaluated using the Beck Depression Scale; quality of life will be evaluated using the SRS-22; and motor imagery will be evaluated.

ability will be evaluated using the Turkish version of the Movement Visualisation Questionnaire-3 (MIQ-3). SPSS (Statistical Package for the Social Sciences) Sciences) statistical program (SPSS 21.0) will be used to analyse the obtained data, with p<0.05 being significant.

DETAILED DESCRIPTION:
The term "posture" is derived from the notion of assuming an upright bodily position, specifically standing. The concept of "body language" refers to the position, alignment, and order of the body parts. The American Academy of Orthopaedic Surgeons (AAOS) defines good posture as a state of muscular and skeletal balance that protects the body from injury and progressive deformities by ensuring that the body structures are aligned in the most appropriate position. Postural disorders are the result of a disruption to this equilibrium. Kyphosis is a prevalent postural issue. A curvature of the thoracic wall that exceeds the standard measurement is referred to as kyphosis. The degree of this curvature of the thoracic wall can be determined by the Cobb angle or kyphosis index. A kyphosis index greater than 13, as determined by the Flexruler, is classified as hyperkyphosis. Thoracic hyperkyphosis is categorised into three distinct types: postural kyphosis, Scheuermann disease, and forms that develop due to congenital deformities. Postural hyperkyphosis is the most prevalent form of kyphosis. Postural hyperkyphosis is characterised by a spinal curvature that occurs in response to external forces, resulting from weakness of the muscles that are effective in the upright position. This curvature of the spine is not rigid, and when patients are asked to stand up straight, the existing curvature can usually be corrected by the patient themselves. Motor imagery (MI) is defined as the visualisation of a movement in the mind without the execution of the movement itself. Research has demonstrated that analogous regions of the brain are stimulated during the process of motor imagery and physical movement. It has been established that individuals can enhance their motor abilities, including lifting weights, playing the piano, and performing surgical procedures, by repeatedly visualising the same movement.The results of this study indicate that motor imagery facilitates motor learning by enhancing synaptic connections in an activity-dependent manner. A review of the extant literature reveals that the participants in studies conducted with healthy individuals are predominantly athletes and musicians. It has been demonstrated that athletes and musicians frequently utilise motor imagery in conjunction with physical training to enhance a variety of skills. The objective of this approach is to enhance performance, alleviate anxiety, and augment body image and self-confidence through its utilisation as a pre-performance rehearsal in athletes. Motor imagery has been demonstrated to be a valuable tool in the domains of motor learning and rehabilitation, particularly in the context of neurological diseases such as stroke, spinal cord injury, and Parkinson's disease. The utilisation of motor imagery in conjunction with physical therapy for stroke patients has been demonstrated to be efficacious in enhancing upper limb function, ambulatory ability, and the patient's capacity to resume daily activities. Despite the paucity of research conducted on individuals with spinal cord injury, it has been posited that motor imagery exerts an indirect influence on motor performance, rather than exerting a direct effect. Instead, it has been hypothesised that motor imagery enhances the function of non-paralyzed muscles. A study conducted on patients suffering from stroke, multiple sclerosis and traumatic brain injury demonstrated that the utilisation of motor imagery in conjunction with physical therapy regimens can yield a favourable impact on functional task performance. In the course of a review of postoperative studies in the literature, Newsome et al. demonstrated the efficacy of motor imagery in reducing the loss of wrist flexion/extension strength that may occur after short-term muscle immobilisation. A number of studies have indicated that motor imagery training in patients who have been immobilised for a short time after anterior cruciate ligament injury is effective in reducing pain, loss of muscle strength, and anxiety, and may improve functional recovery. The preponderance of information regarding motor imagery training has been derived from studies conducted on stroke patients, with a predominant focus on the physical effects of motor imagery training employed in these studies. To the best of the author's knowledge, there have been no studies conducted on the use of motor imagery in the treatment of postural disorders. To date, such studies have been mainly conducted on neurological stroke groups or athletes. Telerehabilitation can be defined as a developing method that aims to provide rehabilitation to patients and clinicians by reducing barriers such as distance, time, and cost using information and communication technology. Telerehabilitation facilitates the provision of rehabilitation services to patients who would otherwise be unable to access them due to geographical, economic or physical limitations. In this context, the objective of the present study was to examine the impact of telerehabilitation motor imagery training on posture, pain, depression, and quality of life, with a view to addressing the existing lacunae in the extant literature on the subject.

ELIGIBILITY:
Inclusion Criteria:

* Having postural kyphosis [Kyphosis index measured with Flexcurve ruler, greater than 13 (35)]
* Having sufficient computer/smartphone usage knowledge to participate in the study or having a relative who can help in this regard
* Having a technological device (computer, mobile phone, tablet) and active internet connection at home
* Being between the ages of 18 and 30

Exclusion Criteria:

* Having a systemic disease
* Being diagnosed with scoliosis
* Having had spinal surgery
* Having a serious cognitive disorder determined by a physician that would prevent the tests

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
THE MOVEMENT IMAGERY QUESTIONNAIRE-3 | Three months
  The Movement Imagery Questionnaire-3 (MIQ-3) consists of 12 items divided into three subscales: Internal Visual Imagery (IVI), External Visual Imagery (EVI), and Kinesthetic Imagery (KI), each containing four items. Responses are rated on a 7-point Likert scale, where 1 indicates "very hard to see/feel" and 7 indicates "very easy to see/feel." For each subscale, the mean score is calculated by summing the scores of its four items and dividing by four, resulting in a value between 1 and 7. Higher scores reflect a greater ease and ability in performing the specific type of imagery. The MIQ-3 has demonstrated good reliability and validity in various languages, including the Turkish version, where Cronbach's alpha values ranged from 0.68 to 0.79 for the subscales and around 0.86-0.87 for the total scale, with test-retest intraclass correlation coefficients between 0.84 and 0.95. This scoring method allows both individual assessment and group-level analysis of imagery ability.
Visual Analog Scale | Three months
  The Visual Analogue Scale (VAS) is a simple, widely used method for measuring subjective experiences such as pain intensity, fatigue, or mood. It typically consists of a 10-centimeter horizontal or vertical line with endpoints labeled to represent the extremes of the sensation being measured, for example, "no pain" at one end and "worst imaginable pain" at the other. Participants are asked to mark a point on the line that best represents their current experience. Higher scores indicate greater intensity of the measured sensation.
New York Posture Rating Scale | Three months
  The New York Posture Rating Scale (NYPRS) is an observational tool used to assess overall body posture by systematically evaluating multiple body segments in both the anterior and lateral views. The scale typically examines areas such as the head, shoulders, spine, hips, knees, and feet, assigning each segment a score based on alignment with an ideal posture. Each body part is scored on a scale, often from 5 (good alignment) to 1 (poor alignment), depending on the degree of deviation from the optimal position. The individual segment scores are then summed to produce a total posture score, with higher totals indicating better postural alignment.
Flexruler Kyphosis Index | Three months
  The Flexicurve (or Flexruler) Kyphosis Index is a clinical method used to quantify the curvature of the thoracic spine, particularly to assess the degree of kyphosis. The procedure involves placing a flexible ruler (Flexicurve) along the contour of the subject's spine while they are standing in a natural posture. Once the ruler has been molded to match the spinal curvature, its shape is traced onto paper. Two key measurements are then taken from the tracing: the length (L), which is the straight-line distance between the starting and ending points of the curve, and the height (H), which is the maximum perpendicular distance from the length line to the deepest point of the curve. The Kyphosis Index (KI) is calculated using the formula:
  KI = (H / L) × 100
  Higher KI values indicate a greater thoracic curvature. This method is simple, inexpensive, and non-invasive, making it useful for both clinical assessment and research, although it measures curvature indirectly and may be less preci

SECONDARY OUTCOMES:
Beck Depression Inventory | Three months
  The Beck Depression Inventory (BDI) is a widely used self-report questionnaire designed to assess the presence and severity of depressive symptoms in adolescents and adults. It consists of 21 items, each addressing a specific symptom or attitude related to depression, such as sadness, pessimism, feelings of guilt, loss of energy, and changes in sleep or appetite. For each item, respondents select one of four statements (scored from 0 to 3) that best describes how they have been feeling over the past two weeks. The total score is obtained by summing the responses to all items, resulting in a range from 0 to 63. Higher scores indicate more severe depressive symptoms. Commonly used severity cut-offs are: 0-9 = minimal depression, 10-18 = mild depression, 19-29 = moderate depression, and 30-63 = severe depression.
SRS-22 (Scoliosis Research Society- 22; SRS-22) | Three months
  The Scoliosis Research Society-22 (SRS-22) questionnaire is a condition-specific, self-reported outcome measure developed to assess health-related quality of life in patients with scoliosis. It contains 22 items divided into five domains: Function/Activity, Pain, Self-Image/Appearance, Mental Health, and Satisfaction with Management. Each item is scored on a 5-point Likert scale, where higher scores indicate better status or greater satisfaction. Domain scores are calculated by averaging the responses to the items within each domain, and the total score is obtained by averaging all domain scores, yielding a range from 1.0 (worst) to 5.0 (best). The SRS-22 is widely used in both clinical practice and research to evaluate the impact of scoliosis and its treatment on patients' daily functioning, emotional well-being, and satisfaction with care. It has been validated in multiple languages and is considered a reliable and sensitive tool for monitoring outcomes over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University- Cerrahpasa, Faculty of Health Science, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No